CLINICAL TRIAL: NCT05655975
Title: The Effect of Gastrojejunostomy Diameters on Weight Loss in Patients Who Underwent Laparoscopic Roux n Y Gastric Bypass
Brief Title: Regain Rate According to gj Anastomosis Size in Gastric Bypass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, Uzman Doktor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ANILERGİNNNN
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Obesity, Morbid; Anastomosis; Roux-en-y Anastomosis Site
Keywords: morbid obesity; Roux n Y gastric bypass; anastomosis diameter; regain; weight loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: All patients undergoing Roux nY gastric bypass will have their anastomotic diameter measured by performing an upper gastrointestinal endoscopy postoperatively. The effect of anastomosis diameter on weight loss will be investigated. All patients will be compared by recording their %EWL, height, weight and BMI values during endoscopy.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The surgeon who will perform the endoscopy after the Roux nY gastric bypass will not know the preoperative body measurements of the patient and the post-operative weight loss, and the patient who has undergone endoscopy will not know the diameter of the gastrojejunostomy anastomosis. Only the person collecting the data of the study will be able to see these results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper gi endoscopy after rygb gastric bypass / weight loss (Active Comparator): In all patients undergoing RYGB gastric bypass and success > %50 EWL , an upper gastrointestinal endoscopy will be performed at the 1st postoperative year to measure the diameter of the gastrojejunostomy anastomosis.
  Interventions: Procedure: upper gi endoscopy
- upper gi endoscopy after rygb gastric bypass / regain (Active Comparator): In all patients undergoing RYGB gastric bypass and regain , an upper gastrointestinal endoscopy will be performed at the 1st postoperative year to measure the diameter of the gastrojejunostomy anastomosis.
  Interventions: Procedure: upper gi endoscopy

INTERVENTIONS:
Procedure: upper gi endoscopy — In all patients undergoing RYGB gastric bypass, an upper gastrointestinal endoscopy will be performed at the 1st postoperative year to measure the diameter of the gastrojejunostomy anastomosis.

SUMMARY:
Obesity has become an important medical and social problem in western countries today. Roux-en-Y gastric bypass (LRYGB) is the most commonly performed surgery for the treatment of morbid obesity in the United States. Recently, there has been a steady increase in the number of surgeons performing bariatric surgery. In 2008, approximately 344,000 bariatric procedures were performed worldwide, of which 220,000 were performed in the United States and Canada. Most of these surgeries were laparoscopic gastric bypass procedures.

There are many technical variations in the performance of the Roux-en-Y gastric bypass, especially when the approach is laparoscopic. Three techniques are commonly used when creating a gastrojejunostomy (GJ): hand-sewn, linear-staple, and circular-staple approaches. The effect of larger-caliber gastrojejunostomy on long-term weight loss is worrisome. Numerous recent reports describe the relationship between gastrojejunostomy enlargement and weight gain after gastric bypass, suggesting that this is a potentially valid concern.

In this study, we aim to determine the effect of this potential GJ enlargement on weight loss.

DETAILED DESCRIPTION:
In this prospective study, 118 patients who underwent laparoscopic Roux-en-Y gastric bypass using linear staples due to morbid obesity at Fatih Sultan Mehmet Training and Research Hospital General Surgery Clinic will be included. The number of samples was calculated by performing impact power analysis. Informed consent form and voluntary consent form will be obtained from all patients.

In our clinic, patients who have undergone LRYGB operation are routinely performed esophagogastroscopy at the end of 1 year, as recommended in the guidelines, to detect any enlargement of the gastric pouch, any ulcers in the anatomical line, or any other pathology. In addition to this process, which is applied as a standard in this study, the measurement of the GJ diameter will be added to the process. In this study, the diameter of the gastrojejunal anastomosis will be measured during the esophago gastroscopy procedure for the patients who applied for the esophagogastroscopy procedure, which we routinely apply to all patients 1 year after the LRYGB operation. This procedure will not incur any additional cost to the routine esophagogastroscopy procedure.

At the end of the procedure, patients will be divided into 2 groups according to their GJ diameters. Those with a GJ diameter of less than 15 mm will be considered as group A, those with a GJ diameter over 15 mm will be considered as group B and evaluated for weight loss. Weight loss will be evaluated as EWL(% excess weight loss) and TWL(% total weight loss). The %TWL variable will be calculated with the formula: [(initial weight - current weight) / (initial weight)] × 100. The %EWL variable will be calculated by the formula: [(initial weight - current weight) / (initial weight - ideal weight)] × 100 The ideal weight for each patient was determined as the weight corresponding to a BMI of 25 kg/m2. The patients will be evaluated in terms of age, gender, comorbidities, preoperative BMI and postoperative BMI.

Esophagogastroscopy procedure: Upper endoscopy will be performed in a medium or deep sedation endoscopy unit. A standard endoscope will be used. The gastric pouch will be measured and examined for ulcers and additional pathologies. The gastrojejunostomy will then be measured using a pre-measured forceps. Patients will be discharged with instructions to maintain an analgesic for pain, proton pump inhibitors, sucralfate, and a clear liquid diet for the first 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone LRYGB operation in the last 15 months in our clinic

Exclusion Criteria:

- Patients who refused to undergo esophagogastroscopy Patients who had another abdominal operation after the operation Patients with gastric ulcer detected during esophagogastroscopy Patients with chronic analgesic use Patients with perioperative complications Patients who did not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
regain by GJ anastomosis | 1 year
  Determination of regain ratio according to anastomosis diameter in the 1st year after RYGB gastric bypass

SECONDARY OUTCOMES:
GJ anastomosis diameter | 1 year
  Finding the average diameter of the gastrojejunostomy anastomosis, which is a critical point in weight loss in RYGB gastric bypass surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Patient information can be shared, especially if requested.